CLINICAL TRIAL: NCT06761638
Title: Comparative Impact of Rhythmic Auditory Stimulation Therapy and Task Specific Training for Improving Motor Functions in Stroke Patients
Brief Title: Comparative Impact of RAST and TST for Improving Motor Functions in Stroke Patients
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall22/760
Record Dates: First submitted 2024-12-26; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rhythmic Auditory Stimulation Therapy (Experimental)
  Interventions: Combination Product: Rhythmic Auditory Stimulation Therapy
- Task-Specific Training (Experimental)
  Interventions: Combination Product: Task-Specific Training

INTERVENTIONS:
Combination Product: Rhythmic Auditory Stimulation Therapy — Rhythmic auditory stimulation (RAS) is a therapeutic technique that uses rhythmic auditory cues, like a metronome or music, to improve motor control and coordination. It is often used in rehabilitation for conditions such as stroke, Parkinson's disease, and other movement disorders to enhance gait and other motor functions through the synchronization of movements to auditory rhythms.
  Arms: Rhythmic Auditory Stimulation Therapy
Combination Product: Task-Specific Training — Task-specific training is a rehabilitation approach that involves practicing specific tasks or activities to improve the performance of those tasks. It is based on the principle that repetitive practice of functional tasks enhances neuroplasticity, leading to better motor skills and functional recovery, especially in stroke and neurological rehabilitation.
  Arms: Task-Specific Training

SUMMARY:
This study evaluates the effectiveness of Rhythmic Auditory Stimulation (RAS) therapy versus Task-Specific Training (TST) in enhancing motor function recovery in stroke patients. RAS uses rhythmic cues to aid movement synchronization, while TST focuses on practicing daily tasks to improve functional ability. In a randomized clinical trial, participants were assigned to either RAS or TST groups, with both receiving structured sessions over several weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients diagnosed with stroke
* Age 40-80 years (46)
* Patients having first ever stroke occurrence
* Moderate motor function impairments (47)
* Patients able to follow instruction

Exclusion Criteria:

* Patients with severe motor impairments
* Patients who had cognitive impairments
* Patients having other neurological conditions and musculoskeletal disorders
* Patients having history of surgery

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-02-15 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Modified Barthel index | 12 Months
  The Modified Barthel Index (MBI) is a crucial tool for assessing functional independence in activities of daily living (ADLs) among patients, particularly those recovering from stroke or other debilitating conditions. It evaluates 10 key self-care and mobility tasks, including feeding, bathing, grooming, dressing, and mobility. Each task is scored based on the level of assistance required, with total scores ranging from 0 (complete dependence) to 100 (complete independence). Higher scores indicate greater independence.
Goniometer | 12 Months
  A goniometer is an instrument used to measure the angle of joints in the body, typically to assess the range of motion (ROM). It is commonly used in physical therapy, rehabilitation, and orthopedics to evaluate joint function and monitor progress in patients recovering from injury or surgery. Range of motions of upper limb measured through this goniometer."

CONTACTS AND LOCATIONS:
Locations (1):
- Azra Naheed Medical College, Superior University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No